CLINICAL TRIAL: NCT02119403
Title: Safety and Efficacy of Hand Held Nitrous, a Device That Delivers 16 Grams of Nitrous Oxide Over 120 Seconds of Inhalation Time.
Brief Title: Hand Held Nitrous Oxide Delivery Device
Acronym: HHN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Strata Medical Innovations (Industry)
Responsible Party: Principal Investigator, Mark Aldana, President, Strata Medical Innovations
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: smi7531
Record Dates: First submitted 2014-04-11; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Anesthesia
Keywords: Minimal Sedation nitrous oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hand Held NitrousTM (Experimental): There are no other interventions to this device
  Interventions: Other: There are no other inteventions.

INTERVENTIONS:
Other: There are no other inteventions. — This device gives patients the opportunity to receive nitrous oxide where no such opportunity exists. There is no other intervention available that creates immediate short term minimal sedation.

SUMMARY:
To study the safety and efficacy of Hand Held Nitrous. A device that delivers 120 seconds of up to 72% nitrous oxide and ambient air.

DETAILED DESCRIPTION:
This study assesses the Hand Held Nitrous Oxide Deliver Device which is intended to be used in nitrous oxide sedation systems by delivering a limited 16 grams of nitrous oxide over a total of 120 seconds of inhalation time.

The device creates short term minimal sedation by delivering a maximum 72% USP grade nitrous oxide / 28 % ambient air combination which quickly drops to under 33% nitrous oxide / 67% ambient air in 60 seconds and stays steady until all the gas is expelled.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing a painful office procedure or exam

Exclusion Criteria:

* Women that are Pregnant
* Children under three years of age

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
This study measures the types of complications (if any) associated with the use of small set amount of nitrous oxide. | The patient is under observation for the length of the procedure or until baseline parameters are met (under 10 minutes). No followup is required.
  This is a short acting device that delivers a small amount of nitrous oxide. The patient responds quickly and recovers quickly (approximately 6 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Howard Beck, MD, Principal Investigator
Locations (2):
- United States (2):
  - Lubbock Urology, Lubbock, Texas
  - Other Medical Practices, Lubbock, Texas